CLINICAL TRIAL: NCT01236482
Title: Comparing Oxytocin and Oxytocin-ergometrine Combinations for Increasing Uterine Tone in Cesarean Delivery: a Pharmacokinetic-pharmacodynamic Study.
Brief Title: Oxytocin in Cesarean Delivery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Yehuda Ginosar, Hadassah Hebrew University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: oxytocined50-HMO-CTIL
Record Dates: First submitted 2010-09-27; First posted 2010-11-08 (Estimated); Last update posted 2010-11-08 (Estimated); Status verified 2010-09

CONDITIONS: Post Partum Hemorrhage
Keywords: Pregnancy; Postpartum hemorrhage; Uterine tone; Oxytocin; Ergometrine; Pharmacokinetic-pharmacodynamic analysis
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxytocin (Active Comparator)
  Interventions: Drug: Oxytocin versus oxytocin-ergometrine
- Oxytocin - ergometrine (Experimental)
  Interventions: Drug: Oxytocin versus oxytocin-ergometrine

INTERVENTIONS:
Drug: Oxytocin versus oxytocin-ergometrine — Group 1: Oxytocin 0.1 I.U./kg/hr (plain) Group 2: Oxytocin 0.1 I.U./kg/hr with ergometrine 2 mcg/kg/hr co-administered Infusion rates determined to achieve equipotential doses based on an earlier PKPD study

SUMMARY:
In this study the investigators hypothesize that infused combinations of oxytocin and ergometrine will exhibit fewer cardiac and neurological side effects than equipotent infusion of oxytocin alone. In order to perform this study the investigators perform the following steps:

1. The investigators validate a quantitative measure of uterine tone as our primary endpoint.
2. The investigators use this endpoint measure in order to determine equipotential doses of different tocotonic drug regimens, based on the ED50 for each.
3. Using equipontial ratios based on the ED50, the investigators compare hemodynamic and other side effects of these tocotonic drug regimes. Plasma levels of oxytocin will be measured.

DETAILED DESCRIPTION:
Obstetric hemorrhage is associated with severe maternal morbidityש and maternal death. The use of tocotonic drugs following delivery is routine practice as part of the active management of the third stage of labor, to increase uterine tone and reduce blood loss. However, the use of these drugs is not without side effects and complications. Oxytocin causes profound vasodilatation, hypotension and increased cardiac output and has been associated with chest pain, reduced arterial oxygen saturation and ST segment changes on ECG. Ergometrine, on the other hand, causes systemic vasoconstriction and hypertension, and reduced cardiac output. As oxytocin and ergometrine are associated with opposing hemodynamic sequelae, there is a rationale to justify the co-administration of both of these drugs in an attempt to cancel out their side effects.

No clinical studies have attempted to titrate the dose of tocotonic drugs against a quantified measure of uterine tone. As a consequence, comparisons of the hemodynamic side effects of oxytocin and other tocotonic agents (particularly ergometrine) have not been based on a knowledge of equipotential doses, making the rational comparison of side effects impossible.

In this study we hypothesize that infused combinations of oxytocin and ergometrine will exhibit fewer cardiac and neurological side effects than equipotent infusion of oxytocin alone. In order to perform this study we perform the following steps:

1) We validate a quantitative measure of uterine tone as our primary endpoint. 2) We use this endpoint measure in order to determine equipotential doses of different tocotonic drug regimens, based on the ED50 for each. 3) Using equipontial ratios based on the ED50, we compare hemodynamic and other side effects of these tocotonic drug regimes. Plasma levels of oxytocin will be measured to enable pharmacokinetic-pharmacodynamic assessments to be made.

ELIGIBILITY:
Inclusion Criteria:

* 80 healthy women presenting for elective repeat cesarean delivery under regional anesthesia.
* All women are ASA class 1-2, aged 18 - 45, with body weight 60-100 kg.

Exclusion Criteria:

* Obstetric risk factors: Pre-eclampsia, abnormalities of placentation (eg placenta accrete, placenta previa), amnionitis, multiple gestation, preterm delivery (< 37 completed weeks), more than three previous cesarean deliveries, previous history of ante-partum or post-partum hemorrhage.
* Maternal medical risk factors: Chronic hypertension, cardiac disease, intracranial pathology, known allergies to oxytocin or ergometrine, autoimmune disorders, SLE, coagulation defect or anticoagulation therapy, amnionitis.
* Women asking for cord blood donations are not included in this study due to the long elapsed time between delivery and the commencement of oxytocin.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2010-11; Primary Completion 2011-05 (Estimated); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
Uterine tone | Up to 30 minutes
  Uterine tone as measured by tissue durometry

SECONDARY OUTCOMES:
Plasma levels of oxytocin | Up to 30 minutes
Subjective side effects | Up to 120 minutes
  Headache, chest pain, shortness of breath

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Hebrew University Medical Center, Jerusalem, Israel